CLINICAL TRIAL: NCT04094129
Title: Evaluation of the Effect of Probiotic Supplementation on Cognitive, Emotional and Related Status on Alzheimer's Dementia Patients
Brief Title: Evaluation of the Effect of Wismemo on Alzheimer's Dementia Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Couldn't sign the contract
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201801746A3
Record Dates: First submitted 2019-09-04; First posted 2019-09-18 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Dementia; Intestinal microbiota; Chronic inflammation; Probiotics
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects received two placebo sachets per day
  Interventions: Dietary Supplement: Placebo
- Probiotic (Experimental): Subjects received two Wismemo sachets with 1x10^10 cfu/day
  Interventions: Dietary Supplement: Wismemo

INTERVENTIONS:
Dietary Supplement: Wismemo — Multi-strain probiotic supplement includes Lactobacillus reuteri GMNL-89, Lactobacillus paracasei GMNL-133 and Lactobacillus plantarum GMNL-141.
  Other Names: Regular treatment with Wismemo
  Arms: Probiotic
Dietary Supplement: Placebo — placebo
  Other Names: Regular treatment with placebo
  Arms: Placebo

SUMMARY:
The present studies demonstrated that pro-inﬂammation, systemic oxidative stress and dysfunction in the brain-gut microbiota axis were involved in Alzheimer's disease (AD) pathogenesis. These results implied the decreased regulation of inflammation-associated risk and microbiota in AD patients could provide the novel strategies for combating the disease. This study was designed to assess the addition of Wismemo in treatment of cholinesterase inhibitors (such as donepezil, rivastigmine, galantamine) in the AD patients.

DETAILED DESCRIPTION:
Previously studies have shown some probiotics could improve stress-related diseases such as anxiety, autism, depression and schizophrenia might be through regulating brain-gut microbiota axis, pro-inﬂammation and oxidative stress. Although recent clinical study indicated that mix-probiotics (containing Lactobacillus acidophilus, Lactobacillus casei, Bifidobacteria bifidum and Lactobacillus fermentum) consumption could improve the cognitive function of dementia patients.

In this clinical study, whether Genmont specific strain probiotics could improve the clinical syndromes and delay worsens in Alzheimer's dementia patients with regular treatment were clarified. A Randomized, double-blind, placebo-controlled clinical trial would be carried out. AD's patients with regular treatment are additive consumption multi-strain probiotic supplement (Wismemo). Half of participants will receive Wismeno and regular treatment in combination, while the other half will receive placebo and regular treatment in combination. To evaluate of the effect of probiotic supplementation on cognitive, emotional and related status on Alzheimer's dementia patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Alzheimer's Dementia. (According to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association diagnostic criteria (NINCDS-ADRDA) and new criteria and guidelines to diagnose Alzheimer's disease were published in 2011 by the National Institute on Aging and Alzheimer's Association)
2. Subjects with administrating cholinesterase inhibitors, such as donepezil, rivastigmine, galantamine.
3. Subjects in age of 55-95 years old.

Exclusion Criteria:

1. Subjects are mixed dementia and vascular dementia.
2. Administration of probiotic dietary supplement 2 weeks before inclusion expect for yakult or yogurt.
3. Participation in other clinical trials.
4. Subjects with thyroid dysfunction.
5. Subjects are receiving cancer drugs.
6. Subjects are receiving immunosuppressant drugs.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) for efficacy | 0, 3, 6 months
  Change in cognitive status was evaluated using the Mini-Mental State Examination (MMSE). MMSE will be assessed at baseline and after intervention. The maximum score is 30. If the scores are less than 24, it would be assessed to the mild dementia. If the scores are less than 16, it would be assessed to the severe dementia.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory (NPI) for efficacy and quality of life | 0, 3, 6 months
  Change from baseline in scores of psychosocial scale and caregiver distress was evaluated using the neuropsychiatric Inventory (NPI) by 12 items respectively. The 12 items include delusion, fantasy, depression, anxiety, etc., The maximum score of psychosocial scale is 144. The maximum score of caregiver distress is 60. Change in scores of total and each item will be assessed at baseline and after intervention.
Change from baseline in levels of peroxidation and antioxidant profiles (MDA and TAC) | 0 and 6 months
  Serum levels may possibly decrease peroxidation or increase antioxidant effects of probiotics.
Change from baseline in levels of inflammatory markers (IL-10,IL-6, IL-1 beta, TNF-alpha and TGF-beta) | 0 and 6 months
  Serum levels may possibly decrease inflammatory or increase anti-inflammatory effects of probiotics.
Change from baseline in levels of inflammatory markers (hs-CRP) | 0 and 6 months
  Serum levels may possibly decrease inflammatory effects of probiotics.
Change from baseline in levels of blood sugar (HbA1c) | 0 and 6 months
  Serum levels may possibly decrease high blood sugar effect of probiotics.
Change from baseline in levels of insulin resistance profile (FPG, insulin and HOMA-IR) | 0 and 6 months
  Serum levels may possibly decrease insulin resistance effect of probiotics.
Gut microbiota for efficacy | 0 and 6 months
  Stool samples at baseline and after intervention will be collected. Gut microbiota profile will be assessed.
Mini-Nutritional Assessment (MNA) for feasibility and efficacy | 0, 3, 6 months
  Change in Mini-Nutritional Assessment (MNA) MNA will be assessed at baseline and after intervention. The maximum score is 14. If the scores are 12-14, it would be assessed to normal malnutrition. If the scores are less than 12, it would be assessed to have the risk of malnutrition. If the scores are less than 8, it would be assessed to the malnutrition.
Defecation frequency and type for feasibility and efficacy | 0, 3, 6 months
  Change in Defecation frequency and type Defecation frequency and type will be assessed at baseline and after intervention.
Zarit's Caregiver Burden Scale for quality of life | 0, 3, 6 months
  Change in total scores of Zarit's Caregiver Burden Scale will be assessed at baseline and after intervention for caregiver stress. The maximum score is 48. The minimum score is 0. If the scores are 0-10, it would be assessed to no to mild burden. If the scores are 10-20, it would be assessed to mild to moderate burden. If the scores are greater than 20, it would be assessed to high burden.
Brief Symptom Rating Scale for quality of life | 0, 3, 6 months
  Change in total scores of Brief Symptom Rating Scale (BSRS-5) will be assessed at baseline and after intervention for caregiver stress. The maximum score is 24. The minimum score is 0. If the scores are 0-5, it would be assessed to good. If the scores are 6-9, it would be assessed to mild emotional distress. If the scores are 10-14, it would be assessed to moderate emotional distress. If the scores are greater than or equal t 15, it would be assessed to severe emotional distress.
Fatigue scale for quality of life | 0, 3, 6 months
  Change in total scores of Fatigue scale will be assessed at baseline and after intervention for caregiver stress. The maximum score is 63. The minimum score is 9.

OTHER OUTCOMES:
Drug Records for feasibility and efficacy | 0, 3, 6 months
  Drug Records including the dosage and frequency The major drugs including cholinesterase inhibitors, such as donepezil, rivastigmine, galantamine will be assessed at baseline and after intervention.
Adverse Events (AE) for feasibility and safety | 0, 3, 6 months
  Expected AE including constipation, diarrhea, flatulence and others gastrointestinal symptoms, unexpected or suspected adverse reaction will be assessed at baseline and after intervention. The AE will be reported by numbers of participants and ratio with different symptoms. And concern the AE of cholinesterase inhibitors with probiotic.
Change from baseline in levels of complete blood count and white blood cell differential count | 0 and 6 months
  To assess the safety after intervention using blood samples.
Change from baseline in levels of AST and ALT | 0 and 6 months
  To assess the liver toxicity after intervention using blood samples.
Change from baseline in levels of BUN, creatinine, microalbumin, GFR, ACR and urine routine examination | 0 and 6 months
  To assess the kidney toxicity after intervention using blood and urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Ching Chen, M.D., Principal Investigator — Chang Gung Memorial Hospital